CLINICAL TRIAL: NCT04090853
Title: Subject Evaluation of the Efficacy of a 1064 nm Diode Laser, Pulsed Electro-Magnetic Fields and Vacuum Assisted Multipolar Radio Frequency for Non-invasive Contouring of the Abdomen and Flanks
Brief Title: Subject Evaluation of a 1064nm Diode Laser/RF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment and Covid19
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL1119
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Subcutaneous Fat Disorder

STUDY DESIGN:
Intervention Model Description: Single group assessed patient feedback regarding satisfaction post treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patient Treatment Group (Other): Up to three Diode and Radio Frequency treatments and up to three additional radio frequency treatments will be performed per patient at the discretion of the principal investigator. Diode treatments will be spaced six weeks apart while the radio frequency treatments will be spaced between 2-3 weeks apart.
  Interventions: Device: Venus Bliss

INTERVENTIONS:
Device: Venus Bliss — The investigational device (Venus Bliss™) is a non-invasive medical aesthetic device designed for body contouring. The device is comprised of a console, four 1064 nm diode laser applicators (60 mm x 60 mm). A belt is included to allow the operator to secure the laser applicators on the lipolysis treatment area, allowing hands free operation. The device uses vacuum assisted radiofrequency (RF) and PEMF (pulsed electromagnetic field) technology which has been shown in clinical studies to be safe and effective in body circumferential reduction and skin tightening.

SUMMARY:
Open-label, baseline-controlled, multi-center study evaluating a 1064 nm diode laser, pulsed electromagnetic fields and vacuum assisted radio frequency for non-invasive fat reduction of the abdomen and flanks.

DETAILED DESCRIPTION:
The study will enroll up to 200 subjects requesting non-invasive lipolysis of the abdomen and flanks. Each subject will receive up to 3 study treatments of the diode laser and up to 3 treatments of the pulsed electromagnetic fields and vacuum assisted radio frequency study treatments. Subjects will be followed at 24 weeks post diode treatments to observe their satisfaction with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and voluntarily provide written informed consent.
2. Healthy male or female, ≥ 18 years of age seeking treatment for unwanted fat in the flanks and or abdomen
3. BMI score is less than 35.
4. Able and willing to comply with the treatment/follow-up schedule and requirements.
5. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study, and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Pregnant, intending to become pregnant, postpartum or nursing in the last 6 months.
2. Any previous liposuction/lipo-sculpture or any type of surgical procedure in the treatment area in the past 12 months.
3. History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection) or use of immunosuppressive medications, 6 months prior to and during the course of the study.
4. History of hyperlipidemia, diabetes mellitus, hepatitis, blood coagulopathy or excessive bleeding.
5. Use of antiplatelet medications (81 mg acetylsalicylic acid daily permitted), anticoagulants, thrombolytics or anti-inflammatory medications within 2 weeks of treatment.
6. Having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
7. Having a permanent implant in the treatment area such as metal plates or an injected chemical substance such as silicone or parenteral gold therapy (gold sodium thiomalate).
8. Use of medications, herbs, food supplements, and vitamins known to induce photosensitivity to light exposure at the wavelength used or history of photosensitivity disorder.
9. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions including but not limited to open lacerations, abrasions, herpes sores, cold sores, active infections.
10. Tattoos in the treatment area.
11. Poor skin quality (severe laxity).
12. Abdominal wall, muscular abnormality or hernia on physical examination.
13. Use of retinoids such as oral isotretinoin (Accutane™) within the past six months or during course of the study.
14. History of keloid or hypertrophic scar formation or poor wound healing in the treatment area.
15. As per the investigator's discretion, any physical or mental condition which may make it unsafe for the subject to participate.
16. Unable or unlikely to refrain from sun exposure, artificial tanning, including the use of tanning booths, prior to (six weeks) and during the course of the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Patient Overall Satisfaction | Week 26
  Patients rate their satisfaction with treatment outcomes at the final follow up visit using a patient survey by answering 12 questions
Patient Treatment Satisfaction | Week 26
  Patients rate their treatment satisfaction using a 5 point Likert Scale. The Likert scale ranges from 1 = very unsatisfied 2 = unsatisfied 3 = neutral 4 = satisfied 5 = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Iger, Study Director — Venus Concept LTD
Locations (3):
- United States (3):
  - Shah Aesthetic Surgery, Denver, Colorado
  - Medical Management Solutions INC, Foxborough, Massachusetts
  - SRS Dermatology, Woodmere, New York

IPD SHARING:
Plan to Share IPD: No